CLINICAL TRIAL: NCT07315360
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL-COHORT STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY OF PF-07328948 IN ADULTS WITH RENAL IMPAIRMENT AND HEALTHY ADULT PARTICIPANTS WITH NORMAL RENAL FUNCTION
Brief Title: A Study to Learn How the Body Processes the Study Medicine PF-07328948 in People With Reduced Kidney Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4921014; C4921014 (Other: Pfizer)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Renal Impairment; Healthy
Keywords: Healthy Volunteers; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: PF-07328948 participants without renal impairment (Experimental): Participants without renal impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948
- Group 2: PF-07328948 participants with severe renal impairment (Experimental): Participants with severe renal impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948
- Group 3: PF-07328948 participants with moderate renal impairment (Experimental): Participants with moderate renal impairment will receive a single dose of PF-07328948, administered orally as 1 PF-07328948 tablet.
  Interventions: Drug: PF-07328948

INTERVENTIONS:
Drug: PF-07328948 — PF-07328948 , 1 tablet orally, once on Day 1

SUMMARY:
The purpose of this study is to learn how the study medicine PF-07328948 is processed by the body and how safe and tolerable it is in adults with different levels of kidney function.

The study will include participants who:

* Are aged 18 to 80 years.
* Either have normal kidney function or long-term reduced kidney function (moderate or severe).
* Have a BMI (body mass index) of 17.5 to 40 kilogram per meter squared, inclusive, and a total body weight of more than or equal to 45 kilograms or 99 pounds.

All participants will receive a single dose of PF-07328948 as a tablet taken by mouth. Participants will stay at a clinical research unit for about 6 days to receive the study medicine and undergo safety checks. Total participation lasts up to 64 days, including screening, inpatient stay, and a follow-up call.

The study is not randomized or blinded, meaning all participants and study staff know which treatment is being given. Group assignment is based on kidney function tests done during screening. The results will help researchers understand how reduced kidney function affects the way PF-07328948 works in the body.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of nonchildbearing potential, between the ages of 18 and 80 years, at the screening visit.
* BMI of 17.5 to 40.0 kg/m2 (inclusive), and a total body weight ≥45 kg (99 lbs).
* Stable renal function, defined as ≤25% difference between 2 measurements of eGFR.
* Group 1 only: at screening, no clinically relevant abnormalities identified by a detailed medical history, physical exam, including blood pressure and pulse rate measurement, ECG and clinical laboratory tests.
* Group 1 only: normal renal function (mean eGFR ≥90 mL/min) based on an average of measures from the screening visits.
* Groups 2 & 3 only: good general health considered acceptable with the expected health status of individuals with chronic renal impairment.
* Groups 2 & 3 only: chronic renal impairment, defined by the following mean eGFR criteria (based on screening visits):

  * Severe RI: 15 ≤ mean eGFR <30 mL/min, not requiring hemodialysis.
  * Moderate RI: 30 ≤ mean eGFR <60 mL/min.

Exclusion Criteria:

* Any condition possibly affecting drug absorption.
* At screening, a positive result for HIV antibodies.
* History of renal, liver, or heart transplantation.
* Urinary incontinence without catheterization.
* Evidence of a prothrombotic state, including history of deep vein thrombosis, pulmonary embolism, or arterial thrombosis, or known genetic predisposition.
* Use of an investigational product within 30 days or 5 half-lives (whichever longer).
* A positive urine drug test or breath alcohol test at screening or admission to study clinic.
* Group 1 only: evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* Group 1 only: screening ECG demonstrating QTcF interval >450 ms or a QRS interval >120 ms.
* Group 1 only: screening seated systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg
* Group 2 & 3 only: presence of acute renal disease
* Group 2 & 3 only: requiring dialysis or anticipated need for dialysis
* Group 2 & 3 only: listed for solid organ transplantation
* Groups 2 & 3 only: persistent severe, uncontrolled hypertension at screening, admission to study clinic, or pre-dose on Day 1.
* Groups 2 & 3 only: screening ECG demonstrating a QTcF interval >470 ms or a QRS interval >120 ms.
* Groups 2 & 3 only: unstable medical conditions or comorbidities that would interfere with study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Fraction of Unbound Drug in Plasma (Fu) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose on Day 1
  Fu is the fraction of unbound drug in plasma, which is calculated by Cu/C (where Cu represents unbound concentration and C represents total concentration).
Unbound AUCinf (AUCinf,u) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose on Day 1
  AUCinf is the area under the plasma concentration-time profile from time zero extrapolated to infinite time. AUCinf,u is the unbound AUCinf.
Unbound Cmax (Cmax,u) of PF-07328948 | At 0 (prior to dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose on Day 1
  Cmax is the maximum plasma concentration. Cmax,u is the unbound Cmax.

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Day 1 to Day 36

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4921014